CLINICAL TRIAL: NCT05386199
Title: The Role of Serotonin in Respiratory and Circulatory Failure in Intensive Care Patients
Brief Title: The Role of Serotonin in Intensive Care Patients
Acronym: SERO-22
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Morten Rostrup, Senior physician and clinical professor, Department of Acute Medicine, Oslo University Hospital
Other Study IDs: REK366749
Record Dates: First submitted 2022-05-06; First posted 2022-05-23 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Sepsis; Septic Shock; Cardiac Arrest With Successful Resuscitation; Multiple Trauma
Keywords: Serotonin; 5-hydroxytryptamine; 5-HT; 5-hydroxyindoleacetic acid; 5-HIAA; Platelet poor plasma-serotonin; PPP-serotonin
MeSH Terms: conditions — Sepsis; Shock, Septic; Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy controls: Healthy volunteers without conditions altering serotonin content in blood.
- Sepsis group: Patients with sepsis or septic shock admitted to ICU and receiving mechanical ventilation.
- Cardiac arrest group: Patients with cardiac arrest and ROSC admitted to ICU and receiving mechanical ventilation.
- Multiple trauma group: Patients with severe multiple trauma admitted to ICU and receiving mechanical ventilation.
- ICU control group: Patients with isolated neurological disease admitted to ICU and receiving mechanical ventilation.

SUMMARY:
Sepsis, cardiac arrest and multiple trauma are potentially life-threatening conditions and common reasons for intensive care unit (ICU) admission. The aim of this study is to investigate the role of the signaling substance serotonin in blood in these conditions.

ELIGIBILITY:
ICU-PATIENTS

Inclusion criteria:

* Active treatment of sepsis, septic shock, cardiac arrest with ROSC or severe multiple trauma.
* Age over 18 years
* Written consent from the patient or preliminary consent from the next of kin.
* Receiving mechanical ventilator treatment upon inclusion.
* Arterial and central venous cannulas present.

Exclusion criteria:

* Withdrawal of consent
* Serotonergic carcinoid syndrome, short bowel or other considerable comorbidity altering serotonin content in blood.
* Intoxication prior to ICU admission.

HEALTHY CONTROLS

Inclusion criteria:

* Age over 18 years and signed written consent.
* Conformed to diet and activity restrictions.

Exclusion criteria:

* Any acute illness or injury
* Ongoing autoimmune, malignant, infectious, or other inflammatory disease.
* Severe psychiatric disease or drug abuse.
* Use of any medication except oral contraceptives last two weeks.
* Withdrawal of consent.

ICU CONTROLS

Inclusion criteria:

* Status epilepticus, encephalitis, stroke, or other localized neurological disease.
* Age over 18 years
* Written consent from the patient or preliminary consent from the next of kin.
* Receiving mechanical ventilator treatment upon inclusion.
* Arterial and central venous cannulas present.

Exclusion criteria:

* Withdrawal of consent
* Clinical signs of infection with focal symptoms or temperature over 38,0°C.
* Biochemical signs of infection or inflammation with leukocytes > 11 x 10^9/l, CRP > 15 mg/l, or PCT > 0,10 μg/l.
* Respiratory failure with PaO2/FiO2 ratio < 40 kPa.
* Circulatory failure with MAP < 60 or need for pressor treatment prior to sedation.
* Thrombocytopenia or thrombocytosis with platelets < 100 or > 400 x 10^9/l.
* Serotonergic carcinoid syndrome, short bowel or other considerable comorbidity altering serotonin content in blood.
* Extracranial autoimmune or malignant disease.
* Severe psychiatric disease or drug abuse.
* Intoxication or physical trauma prior to ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock, cardiac arrest with ROSC or severe multiple trauma, admitted to ICU and receiving mechanical ventilation will be screened for inclusion. A group of healthy controls will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PPP-serotonin | As soon as possible after ICU admission. No more than 3 days after admission.
  Serotonin in platelet poor plasma

SECONDARY OUTCOMES:
PPP-serotonin | End of first week at ICU, an average of 5 days after admission.
  Serotonin in platelet poor plasma
Platelet serotonin | As soon as possible after ICU admission. No more than 3 days after admission.
  Serotonin in platelets
Platelet serotonin | End of first week at ICU, an average of 5 days after admission.
  Serotonin in platelets

OTHER OUTCOMES:
Plasma 5-HIAA | As soon as possible after ICU admission. No more than 3 days after admission.
  5-hydroxyindoleacetic acid in plasma
Plasma 5-HIAA | End of first week at ICU, an average of 5 days after admission.
  5-hydroxyindoleacetic acid in plasma
Urine 5-HIAA | As soon as possible after ICU admission. No more than 3 days after admission.
  5-hydroxyindoleacetic acid in urine
Urine 5-HIAA | End of first week at ICU, an average of 5 days after admission.
  5-hydroxyindoleacetic acid in urine

CONTACTS AND LOCATIONS:
Overall Officials: Morten Rostrup, MD PhD, Principal Investigator — Oslo University Hospital, University of Oslo
Locations (1):
- Oslo University Hospital Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided